CLINICAL TRIAL: NCT02206113
Title: A Sit-to-Stand Intervention for Allina Health Employees: A Pilot Study
Brief Title: Sit to Stand Intervention for Allina Health Employees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allina Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: 3989-1
Record Dates: First submitted 2014-07-28; First posted 2014-08-01 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Stress; Quality of Life
Keywords: Standing workstation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standing workstation - 16 weeks (Experimental): This arm, Standing workstation - 16 weeks, received the intervention of a standing workstation for 16 weeks. For the first 8 weeks, the participants were instructed how long to stand per hour for an 8 hour shift. The second 8 weeks their use was monitored for sustainability.
  Interventions: Behavioral: Standing workstation
- Standing workstation - second 8 weeks (Active Comparator): This arm, Standing workstation - second 8 weeks, received the intervention of a standing workstation for 8 weeks of the study. For the first 8 weeks, the worked at their normal desks without an intervention. The second 8 weeks they received a standing workstation and their use was monitored.
  Interventions: Behavioral: Standing workstation

INTERVENTIONS:
Behavioral: Standing workstation
  Other Names: Ergotron Workfit-S

SUMMARY:
A 16 week pilot study for Allina call center employees to look at the psychological outcomes and biological markers after an intervention of using a standing work station. There were two groups: group 1 received, and was instructed to use, the standing work station for all 16 weeks, group 2 was a wait-list control group and received, and was instructed to use, the standing work station for the second 8 weeks. Psychological outcomes were measured at weeks 0, 4, 8, 12, and 16. Biological markers were measured at weeks 0, 8, and 16.

ELIGIBILITY:
Inclusion Criteria:

* Allina Health Call Center Employee (75% or higher employee status)
* Aged 18 to 65 years
* Provide written informed consent

Exclusion Criteria:

* Unable to stand for 20 minutes continuously unaided
* Home based employees

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-05; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change in self-reported quality of life | Baseline, week 4, week 8, week 12, week 16
  Change in quality of life will be measured through the administration of the PROMIS-29 questionnaire.

SECONDARY OUTCOMES:
Change in waist circumference | Baseline, Week 8, Week 16
  Waist circumference measured in inches
Change in number of minutes stood per day | Baseline, week 8, week 16
  Participants recorded their number of minutes stood at work daily from baseline through week 16.
Change in self-reported stress | Baseline, week 4, week 8, week 12, week 16
  Change in stress will be measured through the administration of the Perceived Stress Scale (PSS).
Change in health promotion and lifestyle choices | Baseline, week 4, week 8, week 12, week 16
  Change in health promotion and lifestyle choices will be measured through the administration of the Health Promoting Lifestyle Profile Questionnaire (HPLP-II).
Change in workplace productivity | Baseline, week 4, week 8, week 12, week 16
  Change in workplace productivity will be measured through the administration of Workplace Productivity and Activity Impairment (WPAI) questionnaire.
Change in self-reported physical activity levels | Baseline, week 4, week 8, week 12, week 16
  Change in self-reported physical activity levels will be measured through the administration of the International Physical Activity Questionnaire (IPAQ)
Change in Body Mass Index (BMI) | Baseline, Week 8, Week 16
  Change in an individual's BMI after being weighed at baseline, week 8, and week 16.
Change in body fat percentage | Baseline, week 8, week 16
  Change in body fat percentage as measured by a BodPod® Assessment.
Change in resting heart rate | Baseline, week 8, week 16
  Change in resting heart rate from baseline to week 16.
Change in blood pressure (systolic and diastolic) | Baseline, week 8, week 16
  Change in both systolic and diastolic blood pressure from baseline to week 16.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Dusek, PhD, Principal Investigator — Allina Health
Locations (1):
- Allina Health, Minneapolis, Minnesota, United States